CLINICAL TRIAL: NCT00281970
Title: Phase II Trial of Weekly Docetaxel (Taxotere®) and Monthly Cisplatin Chemotherapy as Adjuvant Treatment for Patients With Completely Resected Non-small Cell Lung Cancer
Brief Title: Docetaxel and Cisplatin in Treating Patients With Stage I, Stage II, or Stage III Non-Small Cell Lung Cancer That Has Been Completely Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: J0435; P30CA006973 (NIH); JHOC-J0435; 20040761 (Other: JHM IRB); MSKCC-04039; CDR0000455112 (Other: other)
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2016-10

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Docetaxel; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: cisplatin
Drug: docetaxel
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy drugs after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving docetaxel together with cisplatin works in treating patients with stage I, stage II, or stage III non-small cell lung cancer that has been completely removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy and safety of a new dosing schedule and dosing level of docetaxel and cisplatin with the chemotherapy regimens used in the International Adjuvant Lung Cancer Trial (IALT) in patients with completely resected stage IA-IIIB non-small cell lung cancer.

Secondary

* Explore the relationship of time to recurrence, disease-free survival, and overall survival of these patients with levels of circulating DNA and proteomic analysis of serum.

OUTLINE: This is an open-label study.

Patients receive docetaxel IV over 30 minutes on days 1, 8, and 15 and cisplatin IV over 8 hours on day 15. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically proven non-small cell lung cancer (NSCLC)

  * Stage IA-IIIB disease
* Underwent prior complete surgical resection (R0) no more than 2 months ago
* Eligible for cisplatin-based adjuvant chemotherapy

PATIENT CHARACTERISTICS:

* Karnofsky performance status ≥ 70%
* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 8.0 g/dL
* Platelet count ≥ 100,000/mm^3
* Creatinine clearance > 55 mL/min
* Total bilirubin normal
* Alkaline phosphatase, AST, and ALT must meet 1 of the following criteria:

  * Alkaline phosphatase (AP) normal AND AST and ALT ≤ 5 times upper limit of normal (ULN)
  * AP ≤ 2.5 times ULN AND AST and ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST and ALT normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No peripheral neuropathy > grade 1
* No hearing deficit at baseline, even if it does not require a hearing aid or intervention or interfere with activities of daily life (i.e., CTCAE grade 2 or higher)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior postoperative radiation therapy
* No prior chemotherapy for NSCLC
* No prior docetaxel or cisplatin
* No concurrent prophylactic filgrastim (G-CSF) or pegfilgrastim

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-08; Primary Completion 2007-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Total cisplatin dose

SECONDARY OUTCOMES:
Toxicity
Overall survival
Disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Charles M. Rudin, MD, PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (3):
- United States (3):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Result] Azzoli CG, Krug LM, Miller VA, Rizvi NA, Kris MG, Dunne M, Farmer A, Pizzo B, Tyson L, Seeger T, Coleman B, Moore E, Lastinger L, Venkatraman E, Rudin CM. A phase II tolerability study of cisplatin plus docetaxel as adjuvant chemotherapy for resected non-small cell lung cancer. J Thorac Oncol. 2007 Jul;2(7):638-44. doi: 10.1097/JTO.0b013e318074bbd0. PMID 17607120